CLINICAL TRIAL: NCT01618175
Title: Home Oxygen Treatment of Childhood Acute Bronchiolitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOR0013-12CTIL
Record Dates: First submitted 2012-06-10; First posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-05

CONDITIONS: Bronchiolitis, Viral; Home Nursing
Keywords: Bronchiolitis, Viral; Home oxygen therapy; Home Nursing; Outcome and Process Assessment (Health Care); bronchiolitis severity score
MeSH Terms: conditions — Bronchiolitis, Viral

ARMS (1):
- Home oxygen therapy (Experimental): Infants with acute bronchiolitis of low to moderate severity will be discharged home with supplemental oxygen and monitored by phone calls and home visits.
  Interventions: Device: Home oxygen therapy

INTERVENTIONS:
Device: Home oxygen therapy — Oxygen will be provided using a generator, through nasal prongs at a flow rate up to 1 L/min.
  During home stay the parents will be guided on how to suspect signs of clinical deterioration. General treatment: If oxygen saturation by pulse oximeter is greater than 92%, the oxygen will be reduced by a quarter liter per minute while monitoring for 15 minutes. If oxygen saturation decreased to less than 92% of the child will remain with the best previous oxygen flow until the next visit. Once the child reaches - 0.06 l / min for 15 minutes, he will will be checked back on room air. Cessation of oxygen therapy: when the oxygen saturation remains above 92% on room air. Every day that no home visit was performed a phone call will be done and follow-up questionnaire will be filled daily, including oxygen saturation registration.

SUMMARY:
Background: acute bronchiolitis (AB) is a common reason for hospitalization of infants in all population groups, and is usually due to respiratory syncytial virus (RSV) infection. The main cause for hospitalization is often a need for oxygen, but can also include high fever (with a suspected secondary bacterial infection) or increasing respiratory distress. In a minority of cases (some of which can be identified in advance by defining risk groups) a serious illness may develop, including risk of respiratory failure and death. Most cases will just require supplemental oxygen and suction of secretions from the nose (as listed in the recommendations of the American Academy of Pediatrics - AAP). However, this apparently "simple" treatment still requires continued hospitalization. This results in a sharp increase in bed occupancy in Israeli hospital pediatric departments in the winter months. In recent years two studies from developed countries have been published where safety has been demonstrated for home oxygen treatment for babies with AB. However, feasibility studies have not been published yet, for example for populations living in poor conditions. The General Health Services (Klalit) in Israel provides integrated hospital and community health service to the majority of the population living o in our region, thus presenting an opportunity for optimal interventions related to this disease.

DETAILED DESCRIPTION:
Objective: To develop a model of community based safe handling of AB in various communities in southern Israel.

Methods: A prospective intervention study examining the safety and health expenditures in infants with AB treated first in hospital but then discharged earlier with home oxygen while monitored in the community.

Contribution to the focus areas, and the impact of results on health policy planning: 1) Reducing hospitalization days and general financial savings. 2) Ability to implement these findings to populations with variable socio-economic backgrounds. 3) Prevention of nosocomial infections related morbidity.

Innovation and uniqueness in the study: test of this hypothesis precisely in our region, where populations have different socio-economic backgrounds, will build a model that may be suitable for all levels of society.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 2-24 months, but age postconception of over 44 weeks.
2. Ac. bronchiolitis clinical diagnosis: acute respiratory illness including nasal congestion, coughing and wheezing or crackles simplified, Tachypnea or retractions of the chest.
3. X-ray confirms a viral diagnosis of bronchiolitis
4. First attack of wheezing
5. O2 Saturation < 91% room air while arrival to the ER
6. The baby and his family have a way to return to the ER after discharge
7. The family lives a distance of less than 30 minutes drive from the center of Emergency Medicine
8. The baby lives in an environment with no smoking
9. The baby's family is available by phone
10. The baby's family is ready for continuous monitoring of the baby at home 11th. Disease severity index (RDSS) of < 4 (see definitions)

Exclusion Criteria:

1. Previous morbidity: cardiac, pulmonary, neuromuscular, nutrition (including FTT). And congenital or acquired airway problem.
2. Age since conception is less than -44 weeks.
3. History of apneas
4. Bacterial pneumonia suggested by a localized-focal finding on X-ray
5. Previous wheezing attack
6. O2 Saturation > 92% on room air
7. Family has no transportation available follow-up visits
8. The family lives at a distance greater than 30 minutes drive from the medical facility
9. The baby was treated with steroids for this attack
10. There is no continuous monitoring of the baby at home

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Rate of hospital readmission within 10 days after discharge with home oxygen | Within 10 days from discharge home with O2
  Readmission to the hospital because of (1) increased oxygen requirement (> 1 L\ minute through the nose) to maintain oxygen saturation of> 92%. (2) event of apnea. 3) feeding of less than 50% of normal with clinical evidence of dehydration, (4) the parents or pediatrician wish remove the child from the study.